CLINICAL TRIAL: NCT03407911
Title: Rating Comparative Microbiology of Cell Populations Present Around Teeth Affected by Periodontal Disease and Implants Affected by Peri-implant Disease.
Brief Title: Microbiota Around Periodontal Teeth and Implants Affected by Peri-implant Disease.
Status: Completed | Type: Observational
Sponsor: Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele (Other)
Responsible Party: Principal Investigator, Giovanni Barbagallo, Professor, Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Other Study IDs: Barbagallo Perimplantitis
Record Dates: First submitted 2018-01-17; First posted 2018-01-23 (Actual); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Peri-Implantitis; Periodontal Diseases
Keywords: Peri-implant pocket microbiota; Periodontal pocket microbiota
MeSH Terms: conditions — Peri-Implantitis; Periodontal Diseases

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples Without DNA — gingival crevicular fluid around teeth affected by periodontal disease and implant affected by peri-implant disease. samples obtained by inserting paper cone in periodontal and peri-implant sulcus.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Peri-implant microbiota: Bacterial population in Gingival Intracrevicular fluid harvested with adsorbent paper point
  Interventions: Other: Harvested
- Periodontal pocket microbiota: Bacterial population in Gingival Intracrevicular fluid harvested with adsorbent paper point
  Interventions: Other: Harvested
- healthy teeth: Bacterial population in Gingival Intracrevicular fluid harvested with adsorbent paper point
  Interventions: Other: Harvested

INTERVENTIONS:
Other: Harvested — Metagenomic exam of Gingival crevicular fluid harvested by adsorbent paper point around periodontal teeth and implant affected by peri-implantitis

SUMMARY:
The purpose of the study was to evaluate, from a microbiological point of view, microbiota around teeth and implants in the same patient affected by periodontal disease and peri-implant disease, all compared with a healthy tooth. From the identification of particular bacterial species in the examined sites, it is intended to be traced back to the identification of a clear etiopathogenic process, which may shed light on the similarities and differences between the two diseases. In recognition of these mechanisms, the investigators think to develop new therapeutic strategies for the future.

DETAILED DESCRIPTION:
Harvested via sterile paper points, for endodontic use, the sulcular fluid present around a dental element affected by periodontitis, and, in the same patient, the fluid present inside a peri-implant sulcus of a implant affected periimplantitis. If more implants are considered affected by perimplantitis, partecipant will choose the worst as sample site. The same principle will be followed in the case of the tooth affected by periodontal disease. The samples must be underwent to bacterial genomic meta-analysis for the precise identification of bacterial. For a better comparation of the flora, even a healthy tooth from the same patient will be choose like test site and a gingival crevicular fluide will be harvested on it.

The investigators think that the perfect knowledge of the pathogen species is the starter point from a correct therapeutic strategy. But is really important take in mind the individual characteristcs of oral microflora.

The data to be noted at the outset are:

Signs and symptoms of periodontal disease, with precise framing within the Armitage 1999 Classification, and peri-implant disease. For the aim of the study definition of perimplantitis concern an implant with a 4 mm minimal probing depth with bleeding on probing and or suppuration (BOP and Supp) and radiographic bone loss (BL).

Evidence of BL recorded in order of definition of 8th European Consensus Conference of Periodontology Working group 4: BL > 2 mm from the expected bone level if a preliminary rx was absent; Rx 2-3 times the SD of the measurement record (1-1,5 mm) in case a preliminary rx was present.

1. Detections diagnostic radiographic and pre-intervention performed with parallel technique (CBCT optional).
2. Photographs pre, intra and post op (if present)
3. Follow up to 6 months / 1 year (optional) The study provides a GCF harvested around periodontal and peri-implant sulcus in patients recruited for microbiological investigation. The analyzes of the samples are performed "blind". The Probe used is a UNC15 and only one calibrated clinician perform the probing. The pathogen microflora will be compaired with a healthy tooth microflora harvested around a healthy tooth in the same patient.

Pretreatment of the sample sites in order to avoid contamination of the samples by the supragingival bacterial plaque will proceed as follows:

- 2 days prior to sampling, the patient undergoes professional cleaning cups and brushes with the sole purpose of eliminating subgingival plaque. also we will be provided appropriate oral hygiene instruction with brushing twice / day and use of the other instruments where required.

Sampling procedure: The harvested will be carried out through sterile paper point the extent to tip 30 and ISO taper 4%. The sampling technique will be that shown in the figure and marked with the letter c (intracrevicular deep method) until minimum resistance is felt. Each paper point will remain in place for 5 sec, then it will be readily stored in a special sterile container, stored in a refrigerated and delivered within 60 minutes Institute environment that will carry out the examination. Any harvested that show blood contamination will be excluded from the exam.

Microbiological Protocol

1. Sample collection and DNA isolation For the metagenomic analysis, samples of paper strip / paper point by patients included in the study, they will be eluted overnight in PBS (phosphate buffered saline) at 4 ° C. Subsequently, the samples will be centrifuged at 10,000 rpm for 15 min at 4 ° C. After removal of the paper point, the supernatant will be used for the extraction of DNA using the QIAamp DNA Mini kit . The DNA will be quantified with Qubit® 2.0 Fluorometer (Thermo Fisher) using QUBIT Kit dsDNA HS ASSAY KIT (Life Technologies).
2. Analysis of 16S rRNA - Metagenomics The metagenomic analyzes will be conducted on MiSeq platform Illumina. The gene libraries will be sequenced through the MiSeq v3 reagent kits. The 16S rRNA hypervariable regions will be amplified using a DNA concentration of 5 ng / l with the primers V5-V7.

The libraries will be purified by magnetic beads (AgencourtAmpure XP, Beckman), and the concentration and distribution of the fragments of the libraries will be evaluated on DNA Chip 1000 in the microanalyzer 2100 (Agilent Technologies). The analysis of the sequences (amplicon data sets) and the determination of OTU (OperationalTaxonomicUnits) will be performed by QIIME pipeline using as 16S rRNA gene database Green genes .

Inclusion criteria:

* Assets in service for at least one year without any technical GBR (therefore excluded from the study also post-extraction)
* entered Works on native bone
* Fill out a medical history form and a periodontal board dedicated to the event, as well as a card for the clinician which builds on the work published in J ClinPeriodontol 2012; 39 (Suppl 12): 224-244
* Reporting in the type of system board (optional surgical technique)

Exclusion criteria:

* Patients in subintrant systemic conditions that contraindicate the insertion of implants
* Patients in the last three months, after surgery have taken antibiotics or follow any therapy for the resolution of acute events. The same may qualify for the study later.
* Women who are pregnant or nursing or undergoing hormone therapies

ELIGIBILITY:
Inclusion Criteria:

* Implant in service for at least one year without any technical GBR.
* Only Implant inserted on native bone
* Fill out a medical history form and a periodontal board dedicated to the event

Exclusion Criteria:

* Post-extractive implant
* Patients in subintrant systemic conditions that contraindicate the insertion of implants
* Patients in the last three months have taken antibiotics or follow any therapy for the resolution of acute events.
* Women who are pregnant or nursing or undergoing hormone therapies

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: People who received at least one implant loaded for at least one year and affected by peri-implantitis and contemporary present a periodontal tooth and a healthy tooth in own mouth
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2018-04-01 (Actual); Study Completion 2018-06-01 (Actual)

PRIMARY OUTCOMES:
Peri-implant Microbiota | 1 day
  bacterial population around implant affected by peri-implantitis

SECONDARY OUTCOMES:
Microbiota in Peri-implantitis and periodontal disease | 1 day
  Compare the different microbiota around healthy teeth, periodontal teeth and implant affected by peri-implantitis

CONTACTS AND LOCATIONS:
Overall Officials: Sebastiano Ferlito, Study Chair — Azienda Ospedaliera, Universitaria Policlinico Vittorio Emanuele
Locations (1):
- University School of Dental Medicine, Catania, Italy

IPD SHARING:
Plan to Share IPD: Yes
all data
Supporting Information: Study Protocol, SAP, CSR
Time Frame: starting one month after publication
Access Criteria: Sending an e mail with specific request